CLINICAL TRIAL: NCT04765566
Title: A Retrospective, Multi-Center, Real World Study of the BD Bard FLUENCY® PLUS Vascular Stent Graft in the Treatment of Peripheral Artery Disease
Brief Title: FLUENCY® PLUS in the Treatment of Peripheral Artery Disease
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Other Study IDs: BDPI-20-001
Record Dates: First submitted 2021-02-04; First posted 2021-02-21 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Vascular Diseases, Peripheral
Keywords: Iliac Artery Disease; Vascular Stent Graft
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endovascular revascularization of peripheral arteries — Endovascular revascularization of peripheral arteries involves placement of a self-expanding Nitinol Stent encapsulated with ePTFE in diseased vessel segments

SUMMARY:
This is a retrospective, multi-center study to assess the safety and performance by proactively reviewing pre-existing medical records and imaging of patients who had previous placement of FLUENCY® PLUS Vascular Stent Graft in iliac artery vessel(s) between January 2010 and March 2020.

DETAILED DESCRIPTION:
The purpose of this study is to retrospectively collect and analyze data on the FLUENCY® PLUS Vascular Stent Graft to summarize and describe real-world experience, and long-term data regarding its safety and efficacy and to compare these findings with published data on stent-treatment in iliac artery disease. The present study aims to collect clinical data about FLUENCY® treatment of atherosclerotic disease (stenosis, occlusion, dissection) as well as to explore safety and effectiveness data for off-label use in additional indications in the iliac segment that have been described in the scientific literature (vessel rupture, aneurysm).

ELIGIBILITY:
Inclusion Criteria:

* The FLUENCY® PLUS Vascular Stent Graft implantation procedure was for the purpose of lesions in the iliac arteries.
* The FLUENCY® PLUS Vascular Stent Graft was placed between January 2010 and March 2020.
* Male or female ≥ 18 years old at the time of implantation.
* The subject provides written informed consent. The subject may be enrolled without informed consent for anonymous data collection if the responsible Ethics Committee has waived the requirement due to the retrospective study design, and written documentation about this decision is provided to the Investigator and the Sponsor.

Exclusion Criteria:

* The FLUENCY® PLUS Vascular Stent Graft was implanted in an anatomic location other than iliac arteries.
* Absence of a target lesion (i.e. diseased or damaged artery) in the area covered by the FLUENCY® PLUS Vascular Stent Graft.
* Subjects without any existing follow-up information after hospital discharge (This criterion does not apply to subjects who deceased during implantation/prior to discharge).
* The subject was identified with a medical condition, which, in the opinion of the Investigator, may cause him/her to be noncompliant with the protocol, or confound the data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with iliac artery disease.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Freedom from major complications | 30 days
  Freedom from device- and/or procedure-related death or myocardial infarction (MI), or any Target Lesion Revascularization (TLR), or target limb major amputation (above the ankle) through 30 days following the index procedure.
Target Lesion Revascularization | 12 months
  Target Lesion Revascularization (TLR) through 12-months post-index procedure.

SECONDARY OUTCOMES:
Technical Success | During Procedure
  Proportions of lesions with technical success. Technical success is defined as the successful treatment of the target lesion at the index procedure using the FLUENCY® PLUS Vascular Stent Graft, as reported in the questionnaire by the Investigator.
Procedural Success | From Procedure until patient is discharged from hospital (average of 2 days)
  Proportions of patients with technical success and no peri-procedural complications (death, stroke, myocardial infarction (MI), emergent surgical revascularization, significant distal embolization in target limb, and thrombosis of target vessel) prior to hospital discharge.
Target Lesion Revascularization | 24 months, 36 months, 60 months
  Target Lesion Revascularization (TLR) through 24 (if applicable)-, 36 (if applicable)-, and 60 (if applicable)-months post-index procedure.
Target Vessel Revascularization | 12 months, 24 months, 36 months, 60 months
  Target Vessel Revascularization (TVR) through 12-, 24 (if applicable)-,36 (if applicable) and 60 (if applicable)-months post-index procedure. TVR is defined as the first revascularization procedure (e.g. PTA, stenting, surgical bypass, etc.) in the target vessel segment following the index procedure.
Sustained Clinical Success | 30 days, 12 months, 24 months, 36 months, 60 months
  Proportions of patients with sustained cumulative improvement from baseline value of ≥ 1 Rutherford Category at 30-days and 12-, 24 (if applicable)-, 36 (if applicable) and 60 (if applicable)-months post-index procedure, as determined by the Investigator.
Primary Patency | 12 months, 24 months, 36 months, 60 months
  Primary Patency at 12-, 24 (if applicable)-, 36 (if applicable)- and 60 (if applicable)- months post-index procedure (freedom from TLR and restenosis). Restenosis will be assessed by duplex ultrasonography (DUS) or angiography and is present when the target lesion is determined to have >50% stenosis, as determined by the Investigator.
Puncture site complications | From Procedure until patient is discharged from hospital (average of 2 days)
  Presence of peri procedural complications and/or significant post-operative hematoma at puncture site, as determined by the Investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Halena, Prof., Principal Investigator — Medical University of Gdansk
Locations (6):
- Germany (3):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Regensburg, Regensburg
  - Klinikum Nordoberpfalz AG - Klinikum Weiden, Weiden
- Poland (3):
  - Medical University of Gdańsk, Gdansk
  - Mazowiecki Szpital Specjalistyczny (MSS Ostroleka), Ostrołęka
  - Mazowiecki Szpital Brodnowski, Warsaw

IPD SHARING:
Plan to Share IPD: Undecided